CLINICAL TRIAL: NCT04239625
Title: A Phase 2 Multicenter, Double-Masked, Randomized, Placebo-Controlled Study to Investigate the Long Term Safety, Tolerability, Pharmacokinetics and Effects of ALK-001 on the Progression of Stargardt Disease
Brief Title: Open-Label Extension: Tolerability and Effects of ALK-001 on Stargardt Disease (TEASE)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Alkeus Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALK001-P1002-EXT; R01FD004098 (FDA); R01FD006016 (Other Grant/Funding Number: FDA OOPD); R01FD006316 (FDA)
Record Dates: First submitted 2020-01-11; First posted 2020-01-27 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Stargardt Disease; Stargardt Macular Degeneration; Stargardt Macular Dystrophy; Autosomal Recessive Stargardt Disease 1 (ABCA4-related)
MeSH Terms: conditions — Stargardt Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ALK-001 (Experimental)
  Interventions: Drug: ALK-001

INTERVENTIONS:
Drug: ALK-001 — Oral administration of a pill for up to 24 months
  Other Names: C20-D3-Retinyl Acetate; C20 Deuterated vitamin A

SUMMARY:
The purpose of this open-label, multicenter study is to determine the long-term safety, pharmacokinetics and effects of ALK-001 (C20-D3-retinyl acetate) on the progression of Stargardt disease. This study is an extension of NCT02402660 and enrolls participants who are at least 8 years old. Enrollment is by invitation only.

Funding Source - FDA OOPD

ELIGIBILITY:
Simplified Inclusion Criteria:

* Clinical diagnosis of Stargardt disease (STGD1)
* Has at least two ABCA4 disease-causing mutations, unless authorized by sponsor
* Has a best-corrected visual acuity (BCVA) greater than approximately 20/160 in at least one eye
* Healthy as judged by investigator
* Able and willing to comply with study requirements, restrictions and instructions and is likely to complete the 24-month study
* Has been invited to participate in this extension, and has signed and dated the informed consent forms (or assent where appropriate) to participate
* Female of childbearing potential has signed the attestation on contraception requirements

Simplified Exclusion Criteria:

* Is lactating or pregnant
* Has a medical condition likely to prevent compliance with the protocol and/or interfere with absorption of ALK-001 or performance of study procedures
* Has abnormal laboratory result(s) at screening
* Has an ocular disorder that may confound ocular assessments
* Has a history of ocular intervention within 90 days of screening

Ages: 8 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2019-12-20 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability of ALK-001 assessed by incidence and/or clinically-significant changes of a combination of ocular and non-ocular adverse events | From baseline to 24 months
Pharmacokinetic profile of ALK-001 derived from the concentrations of ALK-001 and metabolites in plasma | Up to 24 months

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - Alkeus Site, Phoenix, Arizona
  - Alkeus Site, Los Angeles, California
  - Alkeus Site, Aurora, Colorado
  - Alkeus Site, Gainesville, Florida
  - Alkeus Site, Indianapolis, Indiana
  - Alkeus Site, Grand Rapids, Michigan
  - Alkeus Site, Westbury, New York
  - Alkeus Site, Silverdale, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ma L, Kaufman Y, Zhang J, Washington I. C20-D3-vitamin A slows lipofuscin accumulation and electrophysiological retinal degeneration in a mouse model of Stargardt disease. J Biol Chem. 2011 Mar 11;286(10):7966-7974. doi: 10.1074/jbc.M110.178657. Epub 2010 Dec 14. PMID 21156790
- [Background] Kaufman Y, Ma L, Washington I. Deuterium enrichment of vitamin A at the C20 position slows the formation of detrimental vitamin A dimers in wild-type rodents. J Biol Chem. 2011 Mar 11;286(10):7958-7965. doi: 10.1074/jbc.M110.178640. Epub 2010 Nov 12. PMID 21075840
- [Background] Mihai DM, Jiang H, Blaner WS, Romanov A, Washington I. The retina rapidly incorporates ingested C20-D(3)-vitamin A in a swine model. Mol Vis. 2013 Jul 25;19:1677-83. Print 2013. PMID 23914132
- [Background] Charbel Issa P, Barnard AR, Herrmann P, Washington I, MacLaren RE. Rescue of the Stargardt phenotype in Abca4 knockout mice through inhibition of vitamin A dimerization. Proc Natl Acad Sci U S A. 2015 Jul 7;112(27):8415-20. doi: 10.1073/pnas.1506960112. Epub 2015 Jun 23. PMID 26106163
- [Background] Saad L, Washington I. Can Vitamin A be Improved to Prevent Blindness due to Age-Related Macular Degeneration, Stargardt Disease and Other Retinal Dystrophies? Adv Exp Med Biol. 2016;854:355-61. doi: 10.1007/978-3-319-17121-0_47. PMID 26427432
- See also: Please leave your name if you would like to be contacted to discuss this trial — http://alkeuspharma.com/contact-us/